CLINICAL TRIAL: NCT01162967
Title: PROTOCOL FOR PHASE II CLINICAL TRIAL, RANDOMIZED AND OPEN FOR ETIOLOGICAL TREATMENT OF CHRONIC CHAGAS DISEASE WITH POSACONAZOLE AND BENZNIDAZOLE
Brief Title: Clinical Trial For The Treatment Of Chronic Chagas Disease With Posaconazole And Benznidazole
Acronym: CHAGASAZOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Vall d'Hebron (Other); Tropical Medicine and International Health Unit Drassanes. Barcelona (Unknown); International Health Unit Metropolitana Nord. Santa Coloma. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHAGASAZOL01
Record Dates: First submitted 2010-05-20; First posted 2010-07-15 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole; posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Benznidazole (Active Comparator)
  Interventions: Drug: Benznidazole
- Posaconazole, low dose (Experimental)
  Interventions: Drug: Posaconazole
- Posaconazole, high dose (Experimental)
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Benznidazole — Standard dosage
  Arms: Benznidazole
Drug: Posaconazole
  Arms: Posaconazole, high dose; Posaconazole, low dose

SUMMARY:
The investigators propose the evaluation of posaconazole and benznidazole in humans for the treatment of Chagas disease chronical infection. Exploratory trial of posaconazole antiparasitic activity against Trypanosoma cruzi.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients with serological evidence of Chagas infection and positive PCR real time

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Parasitological cure measured by a real time PCR in blood sample | 12 months after starting treatment
  PCR negative at the end of follow up

SECONDARY OUTCOMES:
Parasitological cure measured by real time PCR in blood sample | End of treatment, weeks 8, 16, 24 and 40 after treatment
  substained parasitological response
Safety and tolerability of both drugs | First 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Molina Israel, MD, Principal Investigator — Infectious Disease Department Vall d'Hebron Hospital; Pahisssa Albert, MD Ph, Study Chair — Infectious Disease Department Vall d'Hebron Hospital; Gomez Jordi, MD, Principal Investigator — International Health Unit Drassanes; Valerio Lluis, MD, Principal Investigator — International Health Unit Metropolitana Nord
Locations (3):
- Spain (3):
  - International Health Unit Metropolitana Nord, Santa Coloma, Barcelona
  - Infectious Disease Department Vall d'Hebron Hospital, Barcelona
  - International Health Unit Drassanes, Barcelona

REFERENCES:
- [Derived] Molina I, Gomez i Prat J, Salvador F, Trevino B, Sulleiro E, Serre N, Pou D, Roure S, Cabezos J, Valerio L, Blanco-Grau A, Sanchez-Montalva A, Vidal X, Pahissa A. Randomized trial of posaconazole and benznidazole for chronic Chagas' disease. N Engl J Med. 2014 May 15;370(20):1899-908. doi: 10.1056/NEJMoa1313122. PMID 24827034